CLINICAL TRIAL: NCT02647697
Title: A Single Oral Dose Study of the Safety, Tolerability, and Pharmacokinetic Profile of Radiprodil in Adult Healthy Volunteers
Brief Title: Study to Evaluate Properties of Radiprodil Given in Oral Solution to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0027; 2015-004376-29 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Volunteers
Keywords: UCB3491; Phase 1; Pharmacokinetics; Radiprodil; Healthy volunteers
MeSH Terms: interventions — radiprodil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiprodil (Experimental): Subjects will receive a single dose of Radiprodil 30 mg in suspension form, orally via a syringe in the morning of Day 1.
  Interventions: Drug: Radiprodil oral

INTERVENTIONS:
Drug: Radiprodil oral — * Active Substance: Radiprodil
  * Pharmaceutical Form: dry granules for oral suspension
  * Concentration: 30 mg
  * Route of Administration: oral use
  Other Names: UCB3491

SUMMARY:
To evaluate the pharmacokinetics (PK) profile of Radiprodil in suspension form in healthy adult subjects.

DETAILED DESCRIPTION:
UP0027 is a Phase 1, single-center, open-label study to investigate the safety, tolerability, and PK profile of radiprodil in healthy adult male and female subjects after a single fasting oral dose of radiprodil 30 mg suspension formulation. A total of 10 subjects will be enrolled in the study.

The primary objective of the study is to evaluate the PK profile of oral radiprodil in suspension form in healthy adult subjects.

The secondary objective of the study is to evaluate the safety and tolerability of oral radiprodil in suspension form in healthy adult subjects.

The exploratory objectives of the study are to evaluate the comparative PK profile of radiprodil from samples collected using 2 alternative microsampling techniques (MITRA™ and Drummond capillary tubes) with that of conventional venous blood samples, and to test the perception of the taste and texture of the oral radiprodil suspension.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, ≥ 18 years to ≤ 45 years of age
* Subject smokes < 10 cigarettes per day and has a score of < 4 on the Fagerström Test for Nicotine Dependence (Heatherthon et al., 1991). The Fagerström Test is not required for nonsmokers (ie, no smoking for at least 6 months)
* Subject has a body mass index (BMI) of 18 to 30 kg/m² (inclusive), with a body weight of at least 50 kg (male) or 45 kg (female)
* Subject has a blood pressure and pulse rate within the normal range in supine position after 5 minutes rest (systolic blood pressure: 90 mmHg to 140 mm Hg, diastolic blood pressure: 45 mmHg to 90 mmHg, pulse rate: 45 bpm to 90 bpm)

Exclusion Criteria:

* Subject has a known hypersensitivity to any components of Radiprodil liquid formulation including the excipients or a history of drug or other allergy that, in the opinion of the Investigator or UCB Study Physician, contraindicates his/her participation
* Subject has received prescription or nonprescription medicines (including over-the-counter medicines and herbal and dietary supplements [including St John's Wort]) within 14 days. Exceptions:

  * Paracetamol for the treatment of mild symptoms (eg, headache or other pain), given at most every 6 h to 8 h, not exceeding 2 g/day, and with a total of no more than 5 g over 7 days
  * Inhaled corticosteroids for seasonal rhinitis
  * Vitamins within recommended daily dose Limits
* Subject has consumed any grapefruit, grapefruit juice, grapefruit-containing products, or star fruit within 14 days prior to administration of Radiprodil
* Subject has a history of unexplained syncope or a family history of sudden death due to long QT syndrome

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The area under the concentration-time curve of Radiprodil from dosing to time t (AUC(0-t)) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
  The area under the concentration-time curve of Radiprodil from dosing to time t (AUC(0-t)) is computed from plasma concentrations of pharmacokinetic samples taken predose and 0.5h, 1h, 1.5h, 2 h, 2.5h, 3 h, 3.5h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose using non-compartmental analysis.
The apparent terminal elimination half-life of Radiprodil (t1/2) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
The maximum observed plasma concentration of Radiprodil (Cmax) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
  The Cmax is the maximum plasma concentration of radiprodil observed from pharmacokinetic samples taken predose and 0.5h, 1h, 1.5h, 2 h, 2.5h, 3 h, 3.5h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
The time of occurrence of Cmax of Radiprodil (Tmax) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
  Time to reach maximum plasma concentration.
The volume of distribution of Radiprodil (Vd) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
The area under the concentration-time curve from dosing extrapolated to infinity of Radiprodil (AUC) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
  The area under the concentration-time curve of Radiprodil from dosing extrapolated to infinity (AUC) is computed from plasma concentrations of pharmacokinetic samples taken predose and 0.5h, 1h, 1.5h, 2 h, 2.5h, 3 h, 3.5h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose dose using non-compartmental analysis.
The individual estimate of the terminal elimination rate constant of Radiprodil (λz) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose
The apparent total body clearance of Radiprodil (CL/F) | Blood samples will be taken pre-dose on Day 1 and 0.5 h, 1 h, Pre-dose, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 3.5 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, and 48 h post dose

SECONDARY OUTCOMES:
Number of subjects reporting at least one treatment-emergent Adverse Event (AE) during the study | From Day 1 to Day 15
  Treatment-emergent adverse event is an adverse event starting after the first study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Up002700001, Groningen, Netherlands

REFERENCES:
- [Derived] Sciberras D, Otoul C, Lurquin F, Smeraglia J, Lappert A, De Bruyn S, Jaap van Lier J. A pharmacokinetic study of radiprodil oral suspension in healthy adults comparing conventional venous blood sampling with two microsampling techniques. Pharmacol Res Perspect. 2019 Jan 28;7(1):e00459. doi: 10.1002/prp2.459. eCollection 2019 Feb. PMID 30705758